CLINICAL TRIAL: NCT05899543
Title: Exploring Patient Experiences of Individuals Joining Chronic Lymphocytic Leukemia Clinical Trials
Brief Title: Determining Clinical Study Experiences of Chronic Lymphocytic Leukemia Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83115421
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research study aims to address the limited understanding of the challenges faced by specific demographic groups of chronic lymphocytic leukemia patients in their participation in clinical trials.

This trial will scrutinize the experiences of patients diagnosed with chronic lymphocytic leukemia as they take part in a separate medical intervention clinical trial. The focus will be on tracking the rates of completion and withdrawal among these individuals.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future chronic lymphocytic leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with chronic lymphocytic leukemia
* Patient is a minimum of 18 years or older
* Able to comprehend the investigational nature of the protocol and provide informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Patients who are currently receiving any other investigational drug
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic lymphocytic leukemia patients who are actively participating in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of chronic lymphocytic leukemia patients who decide to join in a clinical study | 3 months
Rate of patients who remain in an chronic lymphocytic leukemia clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nabhan C, Rosen ST. Chronic lymphocytic leukemia: a clinical review. JAMA. 2014 Dec 3;312(21):2265-76. doi: 10.1001/jama.2014.14553. PMID 25461996
- [Background] Iskierka-Jazdzewska E, Robak T. Investigational treatments for chronic lymphocytic leukemia: a focus on phase 1 and 2 clinical trials. Expert Opin Investig Drugs. 2020 Jul;29(7):709-722. doi: 10.1080/13543784.2020.1770225. Epub 2020 May 27. PMID 32407139
- [Background] Molica S. The clinical safety of ibrutinib in chronic lymphocytic leukemia. Expert Opin Drug Saf. 2015 Oct;14(10):1621-9. doi: 10.1517/14740338.2015.1084286. Epub 2015 Sep 11. PMID 26359217

DOCUMENTS (1):
  • Informed Consent Form (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT05899543/ICF_000.pdf